CLINICAL TRIAL: NCT04880941
Title: The Effect of Progressive Relaxation Exercise Applied to Palliative Caregivers on Coping With Stress and Anxiety Variables
Brief Title: Progressive Relaxation Exercise Applied to Palliative Caregivers on Coping With Stress,Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, PhD., Assistant Prof, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/02
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Palliative Care
Keywords: Progressive Relaxation Exercise; Coping With Stress; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups.
Who Masked: Participant
Masking Description: Progressive Relaxation Exercise and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Relaxation Exercise (Experimental): The Progressive Relaxation Exercise will be held 7 days for 4 weeks, a total of twenty eight sessions. Each session is set as fifty minutes
  Interventions: Behavioral: Progressive Relaxation Exercise
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Behavioral: Progressive Relaxation Exercise — In the progressive relaxation technique, the tension and anxiety in skeletal muscles are relatively relieved.
  Other Names: Control group
  Arms: Progressive Relaxation Exercise

SUMMARY:
It is important to consider the needs of palliative care caregivers and to plan interventions for psychosocial problems.

DETAILED DESCRIPTION:
Cognitive-behavioral methods, which may be applied as relaxation aids in controlling the anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* To be able to communicate adequately
* Not having psychiatric problems
* Volunteering to participate in research
* Caregivers whose patients will be in bed for at least 4 weeks

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Coping With Stress in Palliative Caregivers | 1 week
  Stress Coping Styles Scale-The minimum score to be obtained from the scale is 30, and the maximum score is 120. The high scores indicate that the person copes effectively with stress.
Coping With Stress in Palliative Caregivers | 4 week
  Stress Coping Styles Scale-The minimum score to be obtained from the scale is 30, and the maximum score is 120. The high scores indicate that the person copes effectively with stress.

SECONDARY OUTCOMES:
Anxiety in Palliative Caregivers | 1 week
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety (Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983). It can be used in clinical settings to diagnose anxiety. It also is often used in research as an indicator of caregiver distress. Form Y, its most popular version, has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Anxiety in Palliative Caregivers | 4 week
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety (Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983). It can be used in clinical settings to diagnose anxiety. It also is often used in research as an indicator of caregiver distress. Form Y, its most popular version, has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz ÖZER, PhD, Study Chair — Istanbul Sabahattin Zaim University
Locations (1):
- Istanbul Sabahattin Zain Universitiy, Istanbul, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsitsi T, Charalambous A, Papastavrou E, Raftopoulos V. Effectiveness of a relaxation intervention (progressive muscle relaxation and guided imagery techniques) to reduce anxiety and improve mood of parents of hospitalized children with malignancies: A randomized controlled trial in Republic of Cyprus and Greece. Eur J Oncol Nurs. 2017 Feb;26:9-18. doi: 10.1016/j.ejon.2016.10.007. Epub 2016 Nov 18. PMID 28069156
- [Result] Borji M, Nourmohammadi H, Otaghi M, Salimi AH, Tarjoman A. Positive Effects of Cognitive Behavioral Therapy on Depression, Anxiety and Stress of Family Caregivers of Patients with Prostate Cancer: A Randomized Clinical Trial. Asian Pac J Cancer Prev. 2017 Dec 28;18(12):3207-3212. doi: 10.22034/APJCP.2017.18.12.3207. PMID 29281868
- [Derived] Turan GB, Ozer Z, Demir C. The Effect of Progressive Muscle Relaxation Exercises Applied to Caregivers of Palliative Care Patients on Stress Coping Styles and Anxiety Levels: A Randomised Controlled Trial. Nurs Open. 2025 Feb;12(2):e70149. doi: 10.1002/nop2.70149. PMID 39953943